CLINICAL TRIAL: NCT04693091
Title: A Small-scale Study to Capture Acoustic Pathophysiological Parameters, in the Community, Through a Wearable Device, and to Evaluate the Technical and Practical Feasibility of Utilising This Data as Part of a Medical Device System.
Brief Title: Feasibility of Remote Evaluation and Monitoring of Acoustic Pathophysiological Signals With External Sensor Technology
Acronym: REMAP-WEST-FEA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Senti Tech Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Senti-REMAP-WEST-FEA-1
Record Dates: First submitted 2020-11-15; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Respiratory Disease
Keywords: medical device; remote monitoring
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Intervention Model Description: A pilot stage, exploratory, First-In-Human and traditional feasibility, interventional study of the Senti V1.0 device (CE marked, Class I device), involving 10 patients attending A&E, who are being discharged into the care of the community respiratory team. 5 devices will be used, to cover a range of sizes from extra-small to extra-large.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Senti Arm (Experimental): In stage 1 of this study (6 patients), the patient will apply the device and complete the initial patient survey; questions are around usability, comfort (including feelings of pressure), and acceptability. The Investigator will record the time taken to apply the device. A brief 30 seconds of chest sounds will be recorded from each of the nine sensors on the device in three different settings: standing up, lying down, walking around.
  In stage 2 of this study (10 patients; 6 of whom would be re-recruited from the first stage), the participant will use the device at home over five days. The Investigator will assess the participant daily for any signs of pressure sores or complications from using the device (including topical allergic reactions). The participant will complete a daily survey. The participant is encouraged to remove the device and apply it at their discretion. The participant can opt-out of wearing the device at any stage.
  Interventions: Device: Senti V1.0 Device

INTERVENTIONS:
Device: Senti V1.0 Device — This device class I, CE marked garment, with a similar form to a T-Shirt, embedded with ten sensor modules encased in silicone; the device comes with a charging stand in the form of a clothes hanger. Depending on the outcome of this feasibility study, the device may, in the future, form part of a class IIb medical device system, when accompanied by cloud-based software to listen to both current and historically recorded breath sounds for each Senti patient. The Senti Version One device will be labelled clearly to indicate the device version, on the inside of the garment, conforming to the MDR.
  The garment itself will be made from textile composite, including cotton, elastase, micromodel, spandex, and polyester. All other components (including electronic and other plastic components) will be entirely encased in medical-grade silicone.

SUMMARY:
The aim of this study is to explore the acceptability and feasibility of a novel medical device system for remote monitoring of breath and heart sounds (replicating remotely, and in an easy-to-use garment, that which a clinician would do with their stethoscope to listen to a patient's chest, by evaluating sounds captured through a wearable device (Senti)). As a first-in-man study, the investigators will investigate the safety of the Senti device, the usability and acceptability of the device; and ensure technical and practical feasibility of the device in a real-world clinical setting.

10 patients will be recruited (the study participants) in two tranches (6 and 4) who are being discharged from A&E into the care of the community respiratory team. These patients will wear the Senti device. The first tranche will use the device over a single session lasting 20 minutes only. The second tranche (which will include patients from tranche one, and which will only proceed if no adverse events are detected in tranche one), participants will wear the device at their discretion (particularly encouraged to wear overnight) over the course of 5 days. The investigators will survey the study participants to answer three key questions:

1. What is the feasibility of the Senti data-capture device?
2. Is this device usable in clinical practice?
3. What are the requirements to train patients to use the device?

   The investigators will also consider:
4. Does the device function technically and practically, in real-world clinical scenarios?
5. What are the key expected and unexpected safety issues related to using the device (with a particular emphasis on whether the device is likely to cause pressure sores).

These questions will establish the feasibility of using the Senti data capture device as part of a novel medical device system for the autonomous evaluation and monitoring of bioacoustic signals.

DETAILED DESCRIPTION:
TITLE: Remote Evaluation and Monitoring of Acoustic Pathophysiological parameters with external sensor technology.

DESIGN: First-In-Man and Feasibility study of the Senti Version 1 Device.

AIMS: To explore the acceptability and feasibility of a novel medical device for the remote monitoring and evaluation of acoustic pathophysiological parameters. - To investigate usability and acceptability of the Senti data capture device, and to ensure technical and practical functionality of the device in a real-world clinical scenario.

PRIMARY OUTCOMES: Device feasibility SECONDARY OUTCOMES: Length of time with the device in situ. The ease with which patients can apply the device.

POPULATION ELIGIBILITY: Patients being discharged home with community respiratory team support, after attending A&E.

DURATION: 3 Months. (Recruitment period: 2 months. Analysis and reporting: 1 month).

ELIGIBILITY:
Inclusion Criteria:

* Patients attending A&E who are being discharged from A&E into the care of the community respiratory team.

Exclusion Criteria:

* Patients unable to give their consent.
* Patients with a known sensitivity or allergy to any of the components of the device.
* Patients with any active implanted devices (such as pacemakers or vagal nerve stimulators).
* Patients with existing pressure sores across the area this device would come into contact (predominantly, across the thorax).
* Patients with significant cognitive impairment or limiting physical disabilities - to the extent that they are not able to manage their own ADLs; except where sufficient family or care support is available to manage the device functions (in which case, the device may be used with caution).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Patient-rated device acceptability | 1 month
  Patient questionnaire "on a scale of 1 ("I would not approve at all") to 5 ("I would greatly approve and would like this to become standard practice"), to what extent would you approve of this device being used to enable clinicians to assess your heart and lung sounds as part of a telephone consultation?"
Patient-rated device comfort | 1 month
  Patient questionnaire "on a scale of 1 ("Very difficult to use") to 5 ("Very easy to use"), how easy to use is the device?"
Patient-rated device ease of use | 1 month
  Patient questionnaire "on a scale of 1 ("Too uncomfortable to use for more than an hours or so") to 5 ("As comfortable as a T-Shirt"), how comfortable is the device?"
Expert-rated device data quality | 1 month
  An appropriately qualified person (with clinical experience of auscultation) to rate quality of data captured by the device, as compared subjectively against the quality that they typically expect from standard auscultation, on a scale of 1 ("Much poorer data quality [than standard auscultation]") to 3 ("equivocal data quality") to 5 ("Much higher data quality").
Adverse events and adverse device events. | 1 month
  The number of participants experiencing adverse events, both arising from use of the device or otherwise, will be reported. Adverse events will be categorised as unexpected or expected, serious or otherwise, device-related or un-related.

SECONDARY OUTCOMES:
Length of time spent with the device on the patient. | 1 month
  Length of time over which a patient has used the device, as measured using a structured, binned multiple-choice survey. This is a custom-made scale titled "In the past 24 hours, for how many hours have you worn the Senti device?" with a minimum value of 0 hours and a maximum value of 24 hours. 8 options which include a range of times are available for selection.
Length of time taken for the patient to apply the device | 1 month
  Length of time taken for the patient to put the device on, as measured by an investigator with a stop watch.
Time spent to train patients to use the device. | 1 month
  Length of time taken to train patients to use the device, as measured by an investigator with a stop watch.
Pressure sore EPUAP grade | Through study completion, once per day.
  For those patients who develop pressure sores, the pressure sore will be graded using the European Pressure Ulcer Advisory Panel grading system from a grade of grade 1 through to grade 4, including unclassified gradings and moisture lesions. (Patients will be graded as "No pressure sores" if there are no pressure sores noted on examination).

CONTACTS AND LOCATIONS:
Locations (1):
- Senti Tech, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No